CLINICAL TRIAL: NCT00060736
Title: The Effects of Acute Withdrawal of Estradiol on Mood Symptoms in Women With Perimenopausal Depression
Brief Title: The Effects of Estrogen Withdrawal on Mood Symptoms in Women
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030175; 03-M-0175
Record Dates: First submitted 2003-05-09; First posted 2003-05-12 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2016-04-27

CONDITIONS: Perimenopausal Depression; Post Menopausal; Healthy; Depression
Keywords: Hormone Replacement; Gonadal Steroids; Estrogen; Major Depression; Minor Depression; Perimenopause; Estradiol; Depression; Perimenopausal Depression
MeSH Terms: conditions — Depression; Depressive Disorder, Major

SUMMARY:
This study evaluates the effects on mood when stopping estrogen replacement therapy.

The purpose of this study is to investigate the effects of estrogen levels on perimenopausal depression. This study will examine short-term withdrawal of estrogen in women whose mood had improved with estrogen therapy.

Perimenopause-related mood disorders cause significant distress in a large number of women. Evidence suggests that estradiol may have beneficial effects in women with perimenopausal depression. However, the effect of declining estradiol secretion during perimenopause has not been fully examined.

Peri- and post-menopausal women who experience a remission of perimenopause-related depression symptoms while on estrogen therapy and a control group of healthy volunteers on hormone replacement therapy (HRT) will be switched from their current form of HRT to estradiol for a 3-week period; volunteers will also complete symptom ratings to confirm the absence of mood symptoms. Participants will then be randomly assigned to either continue estradiol or take a placebo (an inactive pill) for an additional 3 weeks. Mood ratings will be used to determine response to estradiol withdrawal.

...

DETAILED DESCRIPTION:
Perimenopause-related mood disorders cause significant distress to a large number of women. Recent studies have reported the therapeutic benefits of estradiol in women with these mood disorders; however, a relevant pathophysiologic role of declining estradiol secretion during the perimenopause has not been demonstrated. In this protocol we wish to investigate the effects of acute withdrawal of estradiol on mood under placebo controlled conditions. Thus, mood and behavior symptoms may be precipitated by the experimental conditions of this protocol. This protocol will address the following hypothesis: women with a past history of perimenopause-related depression but not women without such a history will experience a recurrence of mood and behavioral symptoms during acute estradiol withdrawal but not during continued estradiol administration. The nature of the relationship between the declining secretion of estradiol and mood in perimenopausal depressed women will be examined as follows: Peri- and postmenopausal women reporting the onset of depression during the perimenopause and who report remission of depressive symptoms on estrogen therapy (ET) will be withdrawn from ET under blinded and placebo-controlled conditions. We will recruit as a comparison group asymptomatic women on hormone replacement and without a history of perimenopause-related depression. During a three week baseline phase, all women will be switched from their current form of hormone replacement therapy to estradiol and will complete symptom ratings to confirm the absence of mood symptoms prior to entry into the study. After the screening, all women will be randomized to receive either estradiol or placebo for an additional three weeks. Comparison of mood ratings during these contrasting treatment conditions will allow us to examine the specific role of estrogen withdrawal in depression that is responsive to ET.

ELIGIBILITY:
* INCLUSION CRITERIA:

All subjects for this protocol will be either self-referred in response to newspaper advertisements or referred by their personal physician. The women participating in this protocol will have previously completed the screening protocol # 88-M-0131 and, therefore, will have had the presence or absence of perimenopausal or menopausal reproductive status evaluated and documented.

1. Women with a past perimenopause-related depression (within 12 years) and whose depression responded to ET will be recruited to participate in this randomized, parallel-design, double-blind, placebo-controlled study. Women with histories of either perimenopausal depression that was not responsive to ET or hormone replacement therapy-induced dysphoria due to either the estrogen or the progesterone components of their hormone replacement will be excluded. The diagnosis of perimenopause-related depression will be based on a history of a past depressive episode (major or minor depression confirmed by Structured Clinical Interview for DSM-IV (SCID) or Schedule of Affective Disorders and Schizophrenia-Lifetime Version (SADS-L), respectively) at midlife in association with menstrual cycle irregularity and the history of remission (also confirmed by SCID or SADS-L) of this depression after ET. Additionally, all women will report that they were placed on HRT for the treatment of perimenopausal symptoms, including depression.
2. Age 45 to 65
3. In good medical health

<TAB>

Women without past perimenopausal depression -

To control for the effects of the hormonal manipulations in this protocol, we will also recruit a group of asymptomatic controls who are either currently on ET or were prescribed ET previously and with no previous history of perimenopause-related depression or HRT-induced dysphoria. Women who participate in this study as the asymptomatic comparison group will meet the following criteria:

1. Women who received hormone therapy (HT) with no previous history of perimenopause-related depression or HT-induced dysphoria
2. No current mood or behavioral problems
3. Age 45 to 65
4. In good medical health

EXCLUSION CRITERIA:

1. past history of severe major depression with suicidal ideation
2. current treatment with antidepressant medications
3. history of ischemic cardiac disease, pulmonary embolism, or thrombophlebitis
4. renal disease
5. hepatic dysfunction
6. women with a history of carcinoma of the breast
7. women with a history of uterine cancer, ill-defined pelvic lesions, particularly undiagnosed ovarian enlargement, undiagnosed vaginal bleeding
8. pregnant women
9. cerebrovascular disease (stroke)
10. recurrent migraine headaches

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-05-05; Study Completion 2016-04-27

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Schmidt, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Rossouw JE, Anderson GL, Prentice RL, LaCroix AZ, Kooperberg C, Stefanick ML, Jackson RD, Beresford SA, Howard BV, Johnson KC, Kotchen JM, Ockene J; Writing Group for the Women's Health Initiative Investigators. Risks and benefits of estrogen plus progestin in healthy postmenopausal women: principal results From the Women's Health Initiative randomized controlled trial. JAMA. 2002 Jul 17;288(3):321-33. doi: 10.1001/jama.288.3.321. PMID 12117397
- [Background] Serin IS, Ozcelik B, Basbug M, Aygen E, Kula M, Erez R. Long-term effects of continuous oral and transdermal estrogen replacement therapy on sex hormone binding globulin and free testosterone levels. Eur J Obstet Gynecol Reprod Biol. 2001 Dec 1;99(2):222-5. doi: 10.1016/s0301-2115(01)00398-0. PMID 11788176
- [Background] Schmidt PJ, Nieman L, Danaceau MA, Tobin MB, Roca CA, Murphy JH, Rubinow DR. Estrogen replacement in perimenopause-related depression: a preliminary report. Am J Obstet Gynecol. 2000 Aug;183(2):414-20. doi: 10.1067/mob.2000.106004. PMID 10942479
- [Derived] Rudzinskas S, Hoffman JF, Martinez P, Rubinow DR, Schmidt PJ, Goldman D. In vitro model of perimenopausal depression implicates steroid metabolic and proinflammatory genes. Mol Psychiatry. 2021 Jul;26(7):3266-3276. doi: 10.1038/s41380-020-00860-x. Epub 2020 Aug 12. PMID 32788687
- [Derived] Schmidt PJ, Ben Dor R, Martinez PE, Guerrieri GM, Harsh VL, Thompson K, Koziol DE, Nieman LK, Rubinow DR. Effects of Estradiol Withdrawal on Mood in Women With Past Perimenopausal Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2015 Jul;72(7):714-26. doi: 10.1001/jamapsychiatry.2015.0111. PMID 26018333